CLINICAL TRIAL: NCT03211819
Title: Esthetic Outcome of Computer-guided Versus Free- Hand Immediate Implant Placement in Fresh Extraction Sockets in Esthetic Zone, a Randomized Clinical Trial.
Brief Title: Computer-guided Versus Free- Hand Immediate Implant Placement
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Kotb, Assisstant Lecturer- Prosthodontic Department- Faculty of Dentistry- Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prosthodontic Department
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Dental Implant
Keywords: immediate; esthetics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: due to the nature of the trial only the outcome assessror will be masked from the intervention or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer guided placement (Experimental): In the test group, the computer guided surgical guide manufactured using zenith 3D printer (Dentis, Daegu, Korea) will be used for implant drilling and placement (s-Clean Tapered Implants, Dentis Co., Ltd., Woram-Dong, Dalseo-Gu, Daegu, South Korea) following the manufacture's instructions.
  Then in implants with primary stability > 35 Ncm2, the final abutment will be placed and any further adjustment would be done immediately in the lab and repositioned in place. Then the vacuum stent will be checked in its place again intraorally, then a chair side tooth coloured autopolymerizing resin (Structur 2 SC / QM,VOCO GmbH, Germany) will be injected into the vacuum sheet corresponding to the implant site to construct the temporary crown.
  Interventions: Procedure: immediate implant placement
- free hand placement (Active Comparator): in the control group, the implant will be placed it the socket using free hand technique and according to the manufacturing instruction's (s-Clean Tapered Implants, Dentis Co., Ltd., Woram-Dong, Dalseo-Gu, Daegu, South Korea) . The implants will be placed guided by the socket of the root. Then in implants with primary stability > 35 Ncm2, the final abutment will be placed and any further adjustment would be done immediately in the lab and repositioned in place. Then the vacuum stent will be checked in its place again intraorally, then a chair side tooth coloured autopolymerizing resin (Structur 2 SC / QM,VOCO GmbH,Germany)will be injected into the vacuum sheet corresponding to the implant site to construct the temporary crown.
  Interventions: Procedure: immediate implant placement

INTERVENTIONS:
Procedure: immediate implant placement — A prophylactic antibiotic(Flumox 500mg, Egyptian Int. Pharmaceutical Industries Co.,A.R.E.) would be given to the patient 3 days prior to the surgery. Then on the day of surgery, (AK) will extract the remaining root or tooth in an atraumatic procedure using lancet, periotome (Nordent Manufacturing Inc. U.S.A), minimal force and rotational movement.
  After extraction the socket will be examined for intact labial and palatal bone using depth probe. If all walls are intact the socket would be eligible for immediate implant placement.

SUMMARY:
Patients with fractured anterior teeth indicated for extraction will be recruited to the study. After Extraction of the tooth the socket will be evaluated and if eligible for immediate implant placement, implants will be placed either by free hand or computer guided technique. The pink esthetic score will be evaluated to be the primary outcome.

DETAILED DESCRIPTION:
After diagnosis and history taking the patient will be informed about the sequences of the trial. If the patient wishes to participate and fulfills the clinical examination inclusion criteria, he/she will be sent to perform a Cone Beam Computer Tomography (CBCT) scan while biting on a cotton roll and placing cotton rolls in the vestibule to separate the teeth of interest from the opposing dentition and lips respectively.

Then the investigator will examine the CBCT to ensure the presence of sufficient labial bone. Only patients with sufficient labial bone (1.5-2 mm) will be included in the study. If the patient has less than 1.5 mm labial bone, he/she won't be eligible for immediate implant placement and would be referred to delayed implant placement.

The eligible patients will be recalled for impression making. The principal investigator will do a vacuum stent (2mm hard) on the obtained study cast for temporary crown fabrication after the surgery. The tooth or root to be extracted will be modified on the cast and an artificial tooth would be placed then the vacuum sheet will be pressed on the cast.

At this appointment (impression making) the patient will choose a sealed envelope containing the allocation either to the computer guided group (test group) or free hand group (control group). The patient's name will be written on the envelope to avoid changing the randomization process.

For the test group, the principal investigator (AK) will do virtual planning using Blue Sky ® implant planning software. Proper implant size and diameter will be used and a virtual surgical guide will be constructed in a Standard Triangulation Language (STL) format and exported to a 3D printing machine for printing. After printing the guide would be rechecked for adaptation on the study cast. A metallic sleeve will be placed and adapted to the surgical guide in the proposed implant site, using adhesive to avoid rotation during surgery.

Surgical procedure:

A prophylactic antibiotic would be given to the patient 3 days prior to the surgery. Then on the day of surgery, (AK) will extract the remaining root or tooth in an atraumatic procedure using lancet, periotome, minimal force and rotational movement.

After extraction the socket will be examined for intact labial and palatal bone using depth probe. If all walls are intact the socket would be eligible for immediate implant placement.

In the test group, the computer guided surgical guide will be used for implant drilling and placement following the manufacture's instructions.

While in the control group, after tooth or root extraction implants will be placed free hand guided by the extraction sockets.

Then in implants with primary stability > 35 Ncm2, the final abutment will be placed and any further adjustment would be done immediately in the lab and re-positioned in place. Then the vacuum stent will be checked in its place again intraorally, then a chair side tooth colored auto-polymerizing resin will be injected into the vacuum sheet corresponding to the implant site to construct the temporary crown.

Then occlusion will be checked in maximum intercuspation and lateral movement to avoid any contact with the opposing during the healing period. The patient will be instructed to avoid eating or incising any hard food in the surgical site for at least two weeks.

After a week the patient will be recalled for inspection and postoperative photos to be taken for outcome assessment for both groups. And finally after a period of 6 months the patient would receive a definitive crown.

ELIGIBILITY:
Inclusion Criteria:

* Patients with teeth or remaining roots indicated for extraction in the esthetic zone and eligible for immediate implant placement

  * Sufficient bone labially (at least 1.5-2 mm) assessed after cone beam computer tomography (CBCT) scan
  * Presence of adequate mesio-distal length between the adjacent natural teeth (at least 7 mm), measured on the study cast
  * No overeruption of the opposing teeth to avoid any premature contact with the temporary crown during the osseointegration period.

Exclusion Criteria:

* Presence of active sings or symptoms of acute infection in the tooth or the remaining root

  * Heavy smokers (more than 2 packs per day)
  * Parafunctional habits (clenching or bruxism) diagnosed by history taking and observation of the occlusal surface of the posterior teeth for wear facets
  * Patients with poor oral hygiene
  * Pregnant women
  * Any systemic condition that may interfere with osseointegration (as uncontrolled diabetes, recent head and neck radiation)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Pink Esthetic Score (PES) | 1 week postoperative to surgery
  a scoring system of five points are to be checked and evaluated where 0=incomplete; 1= partially present; 2= completely present
Pink Esthetic Score (PES) | 1 week postoperative to definitive crown
  a scoring system of five points are to be checked and evaluated where 0=incomplete; 1= partially present; 2= completely present

SECONDARY OUTCOMES:
Gingival recession | 1 week and 6 month postoperatively
  yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arısan, V., Karabuda, C. Z., Mumcu, E. & Özdemir, T. Implant Positioning Errors in Freehand and Computer-Aided Placement Methods: A Single-Blind Clinical Comparative Study. Int. J. Oral Maxillofac. Implants 28, 190-204 (2013). 2. Khzam, N. et al. Systematic Review of Soft Tissue Alterations and Esthetic Outcomes Following Immediate Implant Placement and Restoration of Single Implants in the Anterior Maxilla. J. Periodontol. 86, 1321-30 (2015). 3. SCHROPP, L. & ISIDOR, F. Timing of implant placement relative to tooth extraction. J. Oral Rehabil. 35, 33-43 (2008). 4. Al-Sabbagh, M. & Kutkut, A. Immediate Implant Placement. Dent. Clin. North Am. 59, 73-95 (2015).